CLINICAL TRIAL: NCT05482009
Title: Evidence-based Optimization of Chinese and Western Medicine Differentiation and Treatment Scheme for Angina Pectoris After Coronary Revascularization
Brief Title: Treatment of Angina Pectoris After Coronary Revascularization With Integrated Traditional Chinese and Western Medicine
Status: Completed | Type: Observational
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 002-20190701
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Angina Pectoris
Keywords: Integrated Chinese and Western Medicine Treatment; Comprehensive Treatment
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Strong exposure group of traditional Chinese medicine: receiving traditional Chinese medicine treatment + basic western medicine treatment, the cumulative time of traditional Chinese medicine treatment reaches more than 80% of the total course of treatment
  Interventions: Other: Traditional Chinese Medicine Treatment Combined with Western Medicine Basic Treatment
- Moderate Chinese medicine exposure group: received Chinese medicine treatment + western medicine basic treatment, the cumulative time of Chinese medicine treatment reached 30%-79% of the total course of treatment
  Interventions: Other: Traditional Chinese Medicine Treatment Combined with Western Medicine Basic Treatment
- Weak exposure group of traditional Chinese medicine: receiving traditional Chinese medicine treatment + basic western medicine treatment, the cumulative time of traditional Chinese medicine treatment is less than 30% of the total course of treatment
  Interventions: Other: Traditional Chinese Medicine Treatment Combined with Western Medicine Basic Treatment
- Western medicine group: receive basic western medicine treatment only

INTERVENTIONS:
Other: Traditional Chinese Medicine Treatment Combined with Western Medicine Basic Treatment — The cumulative observation and treatment (including Chinese patent medicine, Chinese medicine decoction, Chinese medicine granule, Chinese medicine injection, and western medicine) were more than 5 months, and the follow-up was 1.5 years.
  Groups: Moderate Chinese medicine exposure group; Strong exposure group of traditional Chinese medicine; Weak exposure group of traditional Chinese medicine

SUMMARY:
This study used a multicenter, prospective cohort study. According to whether they received TCM treatment and the degree of exposure to TCM, the cohorts were divided into strong TCM exposure group, TCM exposure group, weak TCM exposure group and Western medicine exposure group. The first three groups received traditional Chinese medicine treatment combined with western medicine basic treatment, and the cumulative treatment time of traditional Chinese medicine reached 80%, 30%-79% or 30% of the total course of treatment, respectively. The fourth group received basic western medicine treatment alone. Among them, Chinese medicines (including Chinese patent medicines, Chinese medicine decoctions, Chinese medicine granules, and Chinese medicine injections) have been used and/or taken for a total of 5 months;

DETAILED DESCRIPTION:
The purpose of this study was to observe whether the combination of traditional Chinese medicine intervention on the basis of standardized western medicine treatment could further reduce the incidence of cardiovascular events in patients with angina pectoris after coronary revascularization compared with western medicine treatment, and to conduct objective follow-up. Evaluation of integrated Chinese and Western medicine interventions. Clinical efficacy of angina pectoris after coronary revascularization and characteristic advantages of TCM syndrome improvement.

The trial is a multicenter, prospective clinical cohort study design. It is expected that 2,000 subjects will be included, and they will be divided into 4 groups according to whether they receive Chinese medicine treatment and the degree of exposure to Chinese medicine. One group received only western medicine basic treatment, and the other three groups received Chinese medicine treatment combined with western medicine basic treatment (the difference was that the cumulative treatment time of Chinese medicine reached 80%, 30%-79% or 30% of the total course of treatment, respectively). Among them, Chinese medicines (including Chinese patent medicines, Chinese medicine decoctions, Chinese medicine granules, and Chinese medicine injections) have been used and/or taken for 5 months in total.

The duration of treatment (including follow-up) in this trial was 24 months. Study data were recorded at 0, 3, 6, 9, 12, 15, 18, 21, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* ①Age ≥18 years old and ≤85 years old;

  * Patients who have undergone coronary revascularization (including coronary bypass and/or PCI) in the past.

    * Those who participated voluntarily and signed the informed consent form.

Exclusion Criteria:

* ①Incomplete case data, unable to provide original surgical data entry;

  * Patients who meet the diagnostic criteria for coronary heart disease, angina pectoris or myocardial infarction, but have not undergone coronary revascularization or failed surgery;

    * Patients who still need continuous mechanical adjuvant therapy after successful coronary revascularization; ④ Combined with other heart diseases, such as malignant arrhythmia (rapid atrial fibrillation, atrial flutter, paroxysmal ventricular tachycardia), or cardiac insufficiency before and after surgery (cardiac function class IV, NYHA class or Killip class), severe cardiopulmonary insufficiency .

      * Those who have a history of hemorrhagic cerebrovascular accident, or a history of ischemic cerebrovascular accident (including TIA) within half a year; ⑥Mental patients or those who may not be able to cooperate with the program requirements and follow-up procedures due to educational level, language barriers and other reasons.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of MACE | Assess once 24 months after taking medicine
  Major adverse cardiovascular events that may have occurred in subjects were recorded throughout the trial,and assessed 24 months after taking medicine.
Readmission rate | Assess once 24 months after taking medicine
  Readmissions for cardiovascular disease were recorded throughout the trial,and assessed 24 months after taking medicine.

SECONDARY OUTCOMES:
Angina attack frequency scale | 3 months
  Subjects were assessed using the Angina attack frequency scale at months 3, 6, 9, 12, 15, 18, 21, and 24. The minimum value is 0 and the maximum value is 6. Higher scores indicate worse subjects.
Angina Attack Duration scale | 3 months
  Subjects were assessed using the Angina Attack Duration scale at months3, 6, 9, 12, 15, 18, 21, and 24. The minimum value is 0 and the maximum value is 6. Higher scores indicate worse subjects.
Angina Pain scale | 3 months
  Subjects were assessed using the Angina Pain scale at months 3, 6, 9, 12, 15, 18, 21, and 24. The minimum value is 0 and the maximum value is 6. Higher scores indicate worse subjects.
Nitroglycerin Dosage scale | 3 months
  Subjects were assessed using the Nitroglycerin Dosage scale at months 3, 6, 9, 12, 15, 18, 21, and 24. The minimum value is 0 and the maximum value is 6. Higher scores indicate worse subjects.
The Seattle angina questionaire | 3 months
  Subjects were assessed using the Seattle Angina Questionnaire at months 0, 3, 6, 9, 12, 15, 18, 21, and 24. The minimum value is 0 and the maximum value is 100. Higher scores indicate better subjects.
NYHA classification | 3 months
  Subjects were assessed at 0, 3, 6, 9, 12, 15, 18, 21, and 24 months using NYHA classification. Results include grades I, II, III, and IV.Higher Class indicate worse subjects.
Traditional Chinese medicine syndrome rating scale | 3 months
  On the 0th, 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th months, the subjects were evaluated using the TCM syndrome score table, and the evaluation results were judged as markedly effective, effective, ineffective or aggravated.
Patient Health Questionaire-9 scale | 3 months
  On the 0th, 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th months,Subjects were assessed using the Patient Health Questionaire-9 scale with a minimum of 0 and a maximum of 27. Higher scores indicate worse subjects.
Generalized Anxiety Disorder -7 scale | 3 months
  On the 0th, 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th months,Subjects were assessed using theGeneralized Anxiety Disorder -7 scale with a minimum of 0 and a maximum of 21. Higher scores indicate worse subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Wang, master, Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine
Locations (1):
- Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided